Study Protocol Title: The effect of platelet-rich fibrin on sensory deficit following anterior cruciate ligament reconstruction caused by bone-tendon-bone graft harvesting

Clinic for Orthopedic Surgery and Traumatology, University Clinical Center of Serbia

Version 01, 18 September 2020

## **COVER PAGE**

Study Protocol Title: Impact of Platelet-Rich Fibrin on Donor Site Regeneration and Functional Recovery after ACL Reconstruction with BPTB Autograft

Version/Date: Version 01, 18 September 2020

NCT number: Not Available

Study Protocol Title: The effect of platelet-rich fibrin on sensory deficit following anterior cruciate ligament reconstruction caused by bone-tendon-bone graft harvesting

Clinic for Orthopedic Surgery and Traumatology, University Clinical Center of Serbia

Version 01, 18 September 2020

## CONSENT FOR PARTICIPATION IN MONITORING THE EFFECTS OF THERAPY

| Participant's Name: |
|---|
| Participant ID No.: |
| By signing this consent form, I confirm that: |
| • I have received both oral and written information regarding the monitoring of therapy effects, and I have read and understood the information provided. |
| • I have had sufficient time to consider my participation and have been given the opportunity to ask any questions. I confirm that I am satisfied with the answers I received. |
| • I understand that my participation is entirely voluntary and that I am free to withdraw at any time without providing a reason, and without any consequences for my future treatment. |
| • I understand that only qualified medical professionals and clinical staff of the Clinic for Orthopedic Surgery and Traumatology of the University Clinical Center of Serbia may access my medical records as needed to ensure proper monitoring and accurate documentation of therapy effects. All personal data will be treated as STRICTLY CONFIDENTIAL. |
| • I understand that the data collected during my participation in this therapy-effect monitoring process will be entered into a database and analyzed, and that it will be used exclusively for scientific purposes. |
| • I have received one signed and dated copy of this information sheet. |
| • I agree to participate in this clinical monitoring of therapy effects. |
| Physician: Date: |

Study Protocol Title: The effect of platelet-rich fibrin on sensory deficit following anterior cruciate ligament reconstruction caused by bone-tendon-bone graft harvesting

Clinic for Orthopedic Surgery and Traumatology, University Clinical Center of Serbia

| Version 01, 18 September 2020 |
|-------------------------------|
| Signature: |
| Name (printed): |
| Patient: |
| Date: |
| Signature: |
| Name (printed): |